CLINICAL TRIAL: NCT05046197
Title: Evaluating the Integration of the Recommended Summary Plan for Emergency Care and Treatment (ReSPECT) Into Primary Care and Its Impact on Patient Treatment and Care.
Brief Title: Evaluating the Integration of the Recommended Summary Plan for Emergency Care Treatment (ReSPECT) Into Primary Care
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Professor Anne Slowther, Professor Anne-Marie Slowther, University of Warwick
Other Study IDs: SOC18/20-21
Record Dates: First submitted 2021-09-01; First posted 2021-09-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Advance Care Planning
Keywords: Advance care planning; Emergency Care Treatment Plans; Primary Care; Social Attitudes; ReSPECT; Evaluation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Work Package 1 - patients and carers: Qualitative interview of 48 Patients, or their carers where the patient lacks capacity, who have had a ReSPECT form completed in the previous 6 months. To include:
  12 patients living in care homes 12 patients living at home (nearing the end of their life) 12 patients living at home (not nearing the end of their life)
- Work Package 1 - GPs: Qualitative interview of 30 General Practitioners who are involved in the ReSPECT process
- Work Package 1 - Care home managers: Qualitative interview of 24 care home managers.
- Work Package 2 - Focus groups/interviews (Members of the Public): Qualitative interview of 30 members of the public with an interest in healthcare regarding attitudes to the ReSPECT process.
- Work Package 2 - Focus groups/interviews (Health and Social Care Professionals): Qualitative interview of 30 Non-GP Health and Social Care Professionals regarding attitudes to the ReSPECT process.
- Work Package 2 - Focus groups/interviews (Faith Leaders): Qualitative interview of 8 faith leaders regarding attitudes to the ReSPECT process.
- Work Package 2 - Survey (Members of the Public): Survey of 1000 members of the public to measure public awareness and acceptability of emergency care treatment plans
- Work Package 2 - Survey (GPs): Survey of 1000 GPs to measure the views of GPs nationally regarding the use of emergency care treatment plans including ReSPECT, in primary care.
- Work Package 3 - Patient records: Patient records of 413 patients within 12 CCGs in England who have had a ReSPECT form completed in the previous 12 months

SUMMARY:
When a person becomes seriously ill health professionals treating them need to make decisions quickly. They may have limited information about the person's medical history or about their wishes about treatment. To help health care professionals decide what is the best treatment for that person Emergency Care Treatment Plans can be used. These record what the person would or would not want to happen in certain situations.

The plans are usually written by the person's doctor after discussing it with them. One type of plan, called ReSPECT (Recommended Summary Plan for Emergency Care and Treatment) is used in many National Health Service hospitals in the UK. However, it might be better to write these plans when the person is living at home before they are admitted to hospital.

ReSPECT forms are now being used by GPs and other primary care staff in the UK. This project plans to study the ReSPECT process in primary care to determine how, when, and why it is used, and what effect it has on patient treatment and care. It will use a mixture of methods for collecting information. The investigators will interview patients, their families, GPs and care home managers to ask them about their experience of the ReSPECT process.

To get a wider range of views, the investigators will also speak to groups of other health professionals, patient organisations and faith leaders, and carry out national surveys of GPs and the general public. The study will also look how at patient records to see how the ResPECT process makes a difference to decisions about medical treatment when a person is seriously ill. The information from these different methods will be brought together at a stakeholder meeting and will be used to work out how the ReSPECT process can work best to improve patient treatment and care.

DETAILED DESCRIPTION:
This is a mixed methods research project comprised of four work packages. The overall theoretical framework within which the study will be analysed is Normalisation Process Theory (NPT). The investigators wish to investigate to what extent ReSPECT is embedded in routine primary care practice and how it is perceived and enacted by health professionals and patients. NPT characterises a set of mechanisms (coherence, cognitive participation, collective action and reflexive monitoring) that influence the embedding of new interventions or processes into clinical practice. The investigators will ask how do clinicians, patients and their families:

1. conceptualise ReSPECT (coherence)
2. initiate or engage with the process (cognitive participation)
3. use the process and the documentation (collective action)
4. evaluate it, and how does it change behaviour (reflexive monitoring)

Work package one This will take place in GP practices and care homes across three CCG areas of England where ReSPECT has been implemented. The investigators will recruit 12 GP practices across the three areas and two care homes associated with each practice. In each practice the investigators will interview patients, the carers of patients who lack capacity, GPs and other practice staff. The investigators will ask the practice to identify two care homes for which they are the main practice and seek to interview the care home manager or a senior member of staff.

Patient/carer interviews

The investigators will recruit up to 48 patient/carers across all sites (12 practices) equally from three groups, which are people:

1. living in a care home
2. living at home, identified as nearing the end of their life (but not in the final stages of a terminal illness)
3. living at home, not identified as nearing the end of life.

Patients and their carers will be identified and invited by practice staff, or the care homes where patients are resident. In each practice the investigators will seek to recruit patients who have had a ReSPECT form completed in the previous six months, or for patients who lack capacity their primary carer or the person who was involved in completion of the ReSPECT form. Potential participants will be invited to take part in an interview, at which the investigators will ask participants if they would agree to be contacted to take part in a second interview 6 months later.

At the first interview the investigators will ask participants:

* What they understand about the ReSPECT process and form
* Their views on the ReSPECT process, when they consider their ReSPECT form should be reviewed and who should initiate this review
* To describe the ReSPECT process from when it was first considered or mentioned through to completion of the form and any updating of the form
* Thoughts and feelings the process engendered; whether the process changed how they viewed themselves, their health/illness, and the prospect of their death; whether they think it resulted in a change to the care, and treatments they received and how they viewed these; their sense of trust in their clinicians and in the health service more generally including whether they trust that the ReSPECT form will receive attention once completed; how the ReSPECT process could be improved. The investigators will ask whether COVID-19 has had any impact on their thinking about ReSPECT or advance care planning in general.

At the follow up interview the investigators will ask participants about major changes to the patient's life context and health/illness since the first interview, including further experience of the ReSPECT process/review. If they have further experience with ReSPECT the investigators will explore this in a similar way to the first interview and prompt for any differences compared to the first interview. Where participants have experienced illness/treatment events the investigators will explore their perception of any influence during this event. With all participants the investigators will explore whether and how their reflections on the ReSPECT process and its impact have changed and what influenced these changes.

GP interviews, conversations with practice staff, and care home interviews In each practice, the investigators will interview the health professional who completed ReSPECT for patient participants or the GP most closely involved in their care if the form was completed in hospital. The investigators will carry out brief conversations with other members of the practice team, for example practice nurses, practice manager, receptionist, asking them about their awareness/use of ReSPECT, and how the process runs in the practice. The investigators will invite the managers of care homes linked to participating practices to take part in an interview about their general experience of ReSPECT and of how clinical decisions are made for residents with a ReSPECT form.

The investigators will also collect pooled anonymous data on;

* practice population demographics
* number of ReSPECT forms recorded
* for people with ReSPECT form: age; ethnicity; eFrailty index; type of residence (care/nursing home or own home/family home) and where ReSPECT form completed (if recorded).

The investigators will analyse interview data using Framework analysis to identify themes that help us understand how and why implementation of ReSPECT varies, the enablers and obstacles to its implementation, and specific ethical concerns.

Work package two In this work package the investigators will engage the public and health professionals in reflection and debate about the concept and use of Emergency Care Treatment Plans in general and ReSPECT in particular. As the use of ECTPs relates to ethical issues and death, the investigators will engage with representatives of all relevant faith communities. Based on the findings of Work Package 1, the investigators will develop two questionnaire surveys. One for the public, and one for primary and community health care professionals.

There are two research strands in this Work Package 2:

* Focus groups/interviews
* Surveys

Focus Groups

Members of the public with an interest in health care will be recruited through patient support groups and local community groups in each of the three areas in which the study takes place. The investigators will purposively select participants from those people expressing an interest to reflect the sociodemographic and ethnic profile of the community until at least 10 people are willing to participate. Health care professionals will be recruited through local branches of professional organisations and social media. The investigators will select to ensure diversity of professional background. Focus group members will be prompted to discuss the following questions:

* What are the benefits for patients, carers, the health service, and wider society of the implementation of ReSPECT?
* What are the dis-benefits of ReSPECT?
* What gets in the way of implementing ReSPECT in a way that optimises its use and value, including access to forms and transfer between health and social care organisations?
* How can the dis-benefits of ReSPECT, and challenges to its use be mitigated?

Interviews The investigators will interview six faith leaders from across the three study areas selected to reflect a diverse range of faith perspectives. Participants will be asked to consider the same topics as the focus group participants and in addition the investigators will explore how the values embedded in ReSPECT sit with key values of their faith and areas were the faith's teaching supports the premise of ReSPECT or could cause challenges for people following that faith. Data from focus groups and interviews will be analysed using Framework analysis.

Surveys Public survey: The investigators will commission the National Centre for Social Research to include questions in the annual British Social Attitudes Survey (BSA), to be presented to 1000 participants.

GP survey: The investigators will distribute the survey through a monthly online survey of UK GPs. The investigators will refine the questions using think aloud interviews with a small number of GPs and pilot the finalised questions with a sample of GPs prior to distribution. The survey provides data on commissioned questions presented to a regionally representative sample of 1000 GPs including partners, salaried non-principals and locums.

Analysis The investigators will analyse associations between the survey outcomes and covariates such as: age, gender, presence/type of chronic disease, functional status (patients), time in practice and practice size (GPs). The most important outcome is the binary outcome 'whether they would complete an emergency care treatment plan' (for themselves if public survey and for their patients if GP survey) for which the investigators will fit a logistic regression model. T.

Work package three In this work package the investigators will look at the quality of completion of ReSPECT forms in primary care and identify to what extent treatment decisions in an acute or emergency situation reflect the recommendations on a person's ReSPECT form. The method will be a retrospective case analysis of ReSPECT forms and the relevant sections of patients' records.

Due to the challenges to obtaining consent from sufficient patients or their carers to achieve a sample that is not biased and includes patients who are likely to have a ReSPECT form and experience an event where the ReSPECT recommendations would be crucial to guiding treatment decisions, the investigators are seeking Confidentiality Advisory Group approval to access the patient records without consent and to use anonymised records for the analysis. The investigators will, through the practices or the relevant care home, write to all patients (or their carers) who have had a ReSPECT form completed in the previous 12 months with information about the study and provide an opportunity for them to opt out.

The ReSPECT form and print outs of the patient record since ReSPECT form completion including hospital discharge letters and ED correspondence up to six months post ReSPECT completion will be generated by the practice and transferred securely to the study team. All included ReSPECT forms will be reviewed using the evaluation tool that the investigators have developed in the recently completed study of ReSPECT in secondary care to assess quality of completion of each section of the form.

For all included ReSPECT forms the relevant data (treatment recommendations including CPR decision (Part 4 of the ReSPECT form) will be extracted from the form. The corresponding medical record will be reviewed to identify the first hospital admission or significant treatment event (defined as an acute episode requiring a medical treatment decision) since ReSPECT form completion.

The record will be compared with the recommendations in section four of the corresponding ReSPECT form to look for congruence. The primary analysis will be on congruence of free text recommendations and clinical care. The investigators will fit a logistic regression model to the binary primary outcome 'congruency or not between what is stated on the ReSPECT form and what is actually implemented' with covariates such as: age, gender, place of residence, health category and cognitive function.

Work package four The study design includes a work package (WP4) to work with people with a learning disability (LD) to co-produce resources and recommendations for the use of ReSPECT. The work package comprises 5 coproduction workshops with up to 16 people with LD.

They will be iterative, and each workshop will include time/space to collate emerging reflections, recommendations and suggestions regarding ReSPECT. An advisory group of 5 people with LD will be formed. The advisory group will meet 8 times during the project and help to co-design the workshops. Researchers will take notes at reference group meetings and workshops and audio record them for the purpose of supplementing fieldnotes. The supplemented fieldnotes will be analysed in using thematic analysis to record emerging themes and summaries of workshops. These outcomes/messages from each workshop will be discussed, reviewed and refined with the Reference Group and presented at the next workshop together with resources to inform the next workshop activities. The final reference group meeting will consider overall findings from the workshops and the recommendations/resources produced. In addition focus groups with up to 20 carers of people with LD will be carried out to explore their views on the use of emergency care treatment plans. Existing evidence highlights poor health outcomes for people with LD and that their needs often go unmet in emergency situations, therefore this work package explores how ReSPECT can be used with people with LD and their carers.

Work package five In this work package the investigators will synthesis their findings from the previous work packages and present the key findings at a stakeholder conference.

ELIGIBILITY:
WP1:

Inclusion Criteria:

Adult (18 years and over) patients with ReSPECT form completed in previous 6 months Carer/next of kin of adult patients without capacity, associated with the ReSPECT form completion General Practitioners involved in ReSPECT process Nursing and care home managers

Exclusion Criteria:

Patients in final stages of terminal illness (expected to die within next four weeks) Patients currently in hospital

WP2 interviews

Inclusion criteria:

Faith leaders

Exclusion criteria:

None

WP2 surveys

Inclusion criteria:

Members of the public General Practitioners

Exclusion criteria:

None

WP3:

Inclusion criteria:

Adult (18 years and over) patients with a ReSPECT form completed in the previous 12 months

Exclusion criteria:

Patients who opt-out Patients in final stages of terminal illness (expected to die within next four weeks)

WP4:

Members of patient and carer organisations Community and faith groups Relevant professional organisations Policy makers and regulatory bodies Members of the national ReSPECT working group

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: WP1:
  * Patients (Primary Care)
  * General practitioners
  * Care home managers
  WP2 Interviews:
  * Members of the public (Community-based)
  * Faith Leaders (Community-based)
  * Health Care Providers
  WP2 surveys
  * Members of the public (Community-based)
  * General Practioners
  WP3:
  - Patients (Primary Care)
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2021-09-19 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of respondents that would be 'willing' to complete an emergency care treatment plan for themselves (if public survey) and for their patients (if GP survey) compared to those that report that they would be 'unwilling' | Single time point cross-sectional survey during Q4 2021
  Response to survey questionnaire administered as part of WP2
Logistic regression of congruency (Yes/No) between recommendations recorded in the ReSPECT form and actual clinical care. | Ongoing data collection between Q3 2021 and Q1 2022
  Analysis of congruency (yes/no) between the recommendations recorded on the ReSPECT form and the actual clinical care delivered to patients, as recorded on their medical records, via logistic regression.

SECONDARY OUTCOMES:
How willing patients are to complete an emergency care plan on a scale of 0 (unwilling) till 10 (unwilling). | Single time point cross-sectional survey during Q4 2021
  Response to survey questionnaire administered as part of WP2
Logistic regression of congruency (Yes/No) between presence of DNACPR decisions recorded in the ReSPECT form and CPR delivered in actual clinical care, as recorded in the patient's medical record. | Ongoing data collection between Q3 2021 and Q1 2022
  Analysis of congruency (yes/no) between the presence of DNACPR decisions recorded on the ReSPECT form and CPR delivered to patients, as recorded on their medical records, via logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Anne-Marie, PhD, Principal Investigator — University of Warwick
Locations (1):
- University of Warwick, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Slowther AM, Harlock J, Bernstein CJ, Bruce K, Eli K, Huxley CJ, Lovell J, Mann C, Noufaily A, Rees S, Walsh J, Bain C, Blanchard H, Dale J, Gill P, Hawkes CA, Perkins GD, Spencer R, Turner C, Russell AM, Underwood M, Griffiths F. Using the Recommended Summary Plan for Emergency Care and Treatment in Primary Care: a mixed methods study. Health Soc Care Deliv Res. 2024 Oct;12(42):1-155. doi: 10.3310/NVTF7521. PMID 39487818